CLINICAL TRIAL: NCT02026622
Title: Comparative Study of Physiological and Cerebrovascular Reactivity in Depression, at the Three Phases of Emotion
Acronym: EMPHILINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PHAO 2012 - TD / EMPHILINE
Record Dates: First submitted 2013-10-29; First posted 2014-01-03 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2015-08

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; cerebrovascular reactivity; emotional reactivity
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psychometrics; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3 groups of subjects (Other): 3 groups: depressive subjects, subjects remitted from depression and control subjects, with the same interventions.
  psychometric tests, MRI, transcranial doppler and TPI, explicitative interview
  Interventions: Behavioral: psychometric tests; Device: MRI; Device: transcranial doppler and TPI; Behavioral: explicitative interview

INTERVENTIONS:
Behavioral: psychometric tests — NEO-PI, MADRS, MINI depression, MMSE, STAI-E, ERD, Anhedonia
Device: MRI — ASL, rest f-MRI, FLAIR, white matter hyper intensities load
Device: transcranial doppler and TPI — transcranial doppler TPI
  Other Names: Tissue Pulsatility Imaging
Behavioral: explicitative interview

SUMMARY:
The main objective is to compare the physiological reactivity (heart and respiratory rates, galvanic skin response, cerebral perfusion, and startle) in the three phases of emotion between depressive subjects, subjects remitted from depression and control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 55
* Informed consent form signed
* Affiliated to a medical insurance
* visual and hearing abilities suitable for exams
* for the depressive group (group D): major depressive disorder according to the DSM-IV criteria as evaluated by the MINI test and MADRS score ≥22
* for the depressive patients in remission's group (group R) : matched on age, at least 1 history of major depressive disorder in the last 10 years and solved for more than 6 months, and MADRS score < 9
* for the control subjects (group T) : matched on age, no psychiatric history, MADRS score < 9

Exclusion Criteria:

* psychotic disorder, bipolar disorder, addiction, suspected dementia (MMSE<25)
* current betablockers or neuroleptics treatment
* any current organic unstable pathology
* history of serious cardiovascular disease (coronary syndrome, cardiac arrythmia, etc.)
* smoking > 10 PY
* history of serious neurologic disease (stroke, cerebral tumour, serious cranial trauma, headache, ...)
* contra-indication to MRI
* uncorrected vision or audition troubles
* patient under juridic protection
* pregnancy, lactating or female without reliable contraception

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
amplitude variations of heart and respiratory rate, cerebral pulsatility, galvanic skin response and startle as measure of physiological reactivity | one day
  amplitude variations of heart and respiratory rate, cerebral pulsatility, galvanic skin response and startle.

SECONDARY OUTCOMES:
MRI data as measure of cerebral perfusion, volume of leukoaraiosis and default network (fMRI at rest) | one day
  cerebral perfusion measured by MRI (Arterial Spin Labelling) volume of leukoaraiosis default network (fMRI at rest)
ultrasound data of doppler as measure of cerebral pulstility | one day
  doppler index of middle cerebral artery At the same time, heart rate variability and cerebral pulsatility at rest will be collected
score of psychometric tests as measure of emotional state | one day
  MADRS score, ERD score, STAI-E score, anhedonia score, Neo-PI score, and the subjective assessment of emotional arousal (self Manikin assessment).
spontaneous verbal production to emotional pictures and explicitative interviews | one day
  spontaneous verbal production to emotional pictures and explicitative interviews

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Tours, Tours, France

REFERENCES:
- [Result] Siragusa MA, Rufin T, Courtois R, Belzung C, Andersson F, Brizard B, Dujardin PA, Cottier JP, Patat F, Remenieras JP, Gissot V, El-Hage W, Camus V, Desmidt T. Left amygdala volume and brain tissue pulsatility are associated with neuroticism: an MRI and ultrasound study. Brain Imaging Behav. 2021 Jun;15(3):1499-1507. doi: 10.1007/s11682-020-00348-w. PMID 32761564